CLINICAL TRIAL: NCT00710255
Title: Role of Leukotrienes and Adenosine in Hyperpnea-induced Bronchospasm Determined by Dynamic Analysis of Exhaled Breath Condensate.
Brief Title: Role of Leukotrienes and Adenosine in Hyperpnea-induced Bronchospasm
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, David Kaminsky, MD, Professor, University of Vermont
Other Study IDs: CHRMS 08-023; Merck IISP 32710
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Asthma, Exercise Induced
Keywords: Asthma; Exercise induced bronchospasm; Hyperpnea induced bronchospasm; leukotrienes; adenosine; exhaled breath condensate
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthmatics: Asthmatics with exercise induced bronchospasm
  Interventions: Procedure: Hyperpnea challenge

INTERVENTIONS:
Procedure: Hyperpnea challenge — 5 minutes of dry air hyperpnea to induce bronchospasm

SUMMARY:
This research is being conducted to help us better understand what causes exercise induced asthma. The investigators hypothesize that two types of chemicals, cysteinyl leukotrienes and adenosine, play an important role. The investigators will be measuring these chemicals in the exhaled breath of volunteers with exercise induced asthma as they undergo a test to mimic exercise induced asthma. The investigators will determine how the levels of these chemicals change in association with how lung function changes before, during and after an episode of exercise induced asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma
* Age 12-75 yrs
* FEV1 > 70% predicted
* HIB response > 10 %
* No smoking last 6 mo and < 10 pack yrs
* No URI last 4 weeks
* No asthma exacerbation last 4 weks
* Able to withhold SABA > 8 hrs and LABA > 24 hrs

Exclusion Criteria:

* Other lung disease
* Cardiac disease or other condition that would preclude safe participation, on theophylline or leukotriene modifiers

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asthmatics with exercise induced bronchospasm
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in level of cystLTs and adenosine | Before and after hyperpnea challenge

SECONDARY OUTCOMES:
Change in pH of EBC and change in pulmonary function | Before and after hyperpnea challenge

CONTACTS AND LOCATIONS:
Overall Officials: David A. Kaminsky, MD, Principal Investigator — University of Vermont
Locations (1):
- Vermont Lung Center, Colchester, Vermont, United States